CLINICAL TRIAL: NCT00395564
Title: Retrospective Chart Review of Patients Who Have Had an Open, Laparoscopic, Ureteroscopic or Percutaneous Surgery
Brief Title: Chart Review of Those Who Have Had Open, Laparoscopic, Ureteroscopic, or Percutaneous Surgery
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Jaime Landman, Professor and Chairman, University of California, Irvine
Other Study IDs: 2008-6613
Record Dates: First submitted 2006-11-01; First posted 2006-11-03 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Urologic Diseases
Keywords: Urologic Surgery
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigator intends to review retrospective de-identified data of patients who have had Open, Laparoscopic, Ureteroscopic or Percutaneous Urologic Surgery.

DETAILED DESCRIPTION:
The investigator reviews retrospective de-identified data of patients who have had Open, Laparoscopic, Ureteroscopic or Percutaneous Urologic Surgery in order to determine different clinical or operative issues.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had Open, Laparoscopic, Ureteroscopic or Percutaneous Urologic Surgery at UCIMC Department of Urology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those who have urologic conditions that need to be treated with open, laparoscopic, ureteroscopic, or percutaneous urologic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Develop outcome effectiveness for minimally invasive procedures | December 2015

CONTACTS AND LOCATIONS:
Overall Officials: Elspeth McDougall, Principal Investigator — University of California Irvine-Department of Urology
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States